CLINICAL TRIAL: NCT05323851
Title: How Future Surgery Will Benefit From Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Related Measures Perspective From Italian Young Surgeon Society (SPIGC)
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: SPIGC (Unknown)
Responsible Party: Principal Investigator, Roberta Angelico, MD, PhD, FEBS, Senior Lecturer, Department of Surgical Science, Tor Vergata University., University of Rome Tor Vergata
Other Study IDs: COVID-Italiansurg-SPIGC
Record Dates: First submitted 2022-03-30; First posted 2022-04-12 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: COVID-19; Health Behavior
Keywords: COVID-19; Survey; Enhanced Recovery After Surgery (ERAS) protocol; perioperative management
MeSH Terms: conditions — COVID-19; Health Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgeon: Any Resident, Fellow, PhD candidate, consultant or attending surgeon in any surgical specialty in Italy
  Interventions: Behavioral: COVID-surg-SPIGC questionnaire

INTERVENTIONS:
Behavioral: COVID-surg-SPIGC questionnaire — The questionnaire aimed to evaluate how the COVID-19 pandemic determined a shift in daily practice through a multidimensional assessment of surgical clinical care in three different time frames.

SUMMARY:
The coronavirus 2019 pandemic (COVID-19) strongly affected clinical care worldwide. Due to a shortage of hospitals and beds in intensive care units (ICU), in Italy during outbreaks, surgical resources were temporarily and partially shifted to COVID-19 patients. In addition, the risk of cross-infection could have determined a shit in surgical perioperative care.

To counterbalance these limitations, many centers routinely changed their clinical practice, which could be maintained by surgeons across Italy. The aim of the present study is to evaluate how the COVID-19 pandemic determined a change in daily clinical practice among all specialties.

DETAILED DESCRIPTION:
The purpose of this investigation, organized by the Italian Young Surgeon Society (S.P.I.G.C.), is to establish the impact of the coronavirus 2019 pandemic (COVID-19) on clinical care in Italy.

There will be collected from any Italian surgeon (resident, Fellow, Doctor of Philosophy (Ph.D.) candidate, attending surgeon, professor) impressions by completing a survey on this topic.

The analysis is divided into three study periods. For each question, participants must answer for each period. Time frames were divided according to three distinct phases of the pandemic: pre-COVID-19 period, COVID-19 pandemic period, COVID-19 Endemic period.

The pre-COVID-19 period was defined between eighth March 2019 and seventh March 2020, whereas the COVID-19 pandemic period was identified between the declaration of Italian lockdown measures (eighth March 2020) until the release of this questionnaire (sixteenth March 2022) with the periodic pandemic outbreaks. Finally, COVID-19 endemic period was described as a future phase where lockdown measures and social distancing will be removed.

ELIGIBILITY:
Inclusion Criteria:

* Resident, Fellow, PhD candidate, consultant or attending surgeon in Italy in the following surgical specialties: cardiothoracic surgery, colon and rectal surgery, general surgery, gynecology and obstetrics, gynecologic oncology, neurological surgery, ophthalmic surgery, oral and maxillofacial surgery, orthopedic surgery, otorhinolaryngology, pediatric surgery, plastic and maxillofacial surgery, urology, and vascular surgery

Exclusion Criteria:

* undergraduate students
* Non-Surgical consultant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any attending surgeon, resident, PhD candidate, or fellow in any surgical specialty in Italy
Sampling Method: Non-Probability Sample
Enrollment: 581 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
The measure of the Italian surgical daily practice before coronavirus pandemic (COVID-19) | 12 months before the beginning of COVID-19 emergency in Italy (between eighth March 2019 and seventh March 2020)
  Analysis of this outcome will be held through COVID-surg-SPIGC questionnaire. Variables will be collected as absolute numbers (e.g., number of procedures in a month) or percentages (e.g., percentage of elective surgery compared to total procedures).
  A sub-analysis will be held regarding the different surgical subspecialties, Italian medical centers, and academic grades.
The measure of the Italian surgical daily practice during coronavirus pandemic (COVID-19) | COVID-19 pandemic (between eighth March 2020 and sixteenth March 2022)
  Analysis of this outcome will be held through COVID-surg-SPIGC questionnaire. Variables will be collected as absolute numbers (e.g., number of procedures in a month) or percentages (e.g., percentage of elective surgery compared to total procedures).
  A sub-analysis will be held regarding the different surgical subspecialties, Italian medical centers, and academic grades.

OTHER OUTCOMES:
Expectation of the Italian surgical daily practice after coronavirus pandemic (COVID-19) | 12 months after the release of COVID-surg-SPIGC questionnaire.
  Analysis of this outcome will be held through COVID-surg-SPIGC questionnaire. Variables will be collected as absolute numbers (e.g., number of procedures in a month) or percentages (e.g., percentage of elective surgery compared to total procedures).
  A sub-analysis will be held regarding the different surgical subspecialties, Italian medical centers, and academic grades.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Angelico, Principal Investigator — University of Rome Tor Vergata
Locations (3):
- Italy (3):
  - Azienza ospedaliera S. Camillo Forlanini, Roma, Rome
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Università degli Studi di Roma Tor Vergata, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pertile D, Gallo G, Barra F, Pasculli A, Batistotti P, Sparavigna M, Vizzielli G, Soriero D, Graziano G, Di Saverio S, Meniconi RL, Guaitoli E, Mazzarri A; SPIGC Working Group. The impact of COVID-19 pandemic on surgical residency programmes in Italy: a nationwide analysis on behalf of the Italian Polyspecialistic Young Surgeons Society (SPIGC). Updates Surg. 2020 Jun;72(2):269-280. doi: 10.1007/s13304-020-00811-9. Epub 2020 Jun 16. PMID 32557207
- [Background] Vanni G, Legramante JM, Pellicciaro M, DE Carolis G, Cotesta M, Materazzo M, Buonomo C, Farinaccio A, Santori F, Saraceno F, Ielpo B, Aiello F, Paganelli C, Grande M, DE Andreis G, Chiocchi M, Palombi L, Buonomo OC. Effect of Lockdown in Surgical Emergency Accesses: Experience of a COVID-19 Hospital. In Vivo. 2020 Sep-Oct;34(5):3033-3038. doi: 10.21873/invivo.12137. PMID 32871849
- [Background] Buonomo OC, Materazzo M, Pellicciaro M, Caspi J, Piccione E, Vanni G. Tor Vergata University-Hospital in the Beginning of COVID-19-Era: Experience and Recommendation for Breast Cancer Patients. In Vivo. 2020 Jun;34(3 Suppl):1661-1665. doi: 10.21873/invivo.11958. PMID 32503826
- [Background] Ielpo B, Podda M, Pellino G, Pata F, Caruso R, Gravante G, Di Saverio S; ACIE Appy Study Collaborative. Global attitudes in the management of acute appendicitis during COVID-19 pandemic: ACIE Appy Study. Br J Surg. 2021 Jun 22;108(6):717-726. doi: 10.1002/bjs.11999. Epub 2020 Oct 8. PMID 34157090
- [Background] Manzia TM, Angelico R, Toti L, Pisani G, Vita G, Romano F, Pirozzi BM, Vinci D, Cacciola R, Iaria G, Tisone G. The hamletic dilemma of patients waiting for kidney transplantation during the COVID-19 pandemic: To accept or not to accept (an organ offer)? Transpl Infect Dis. 2021 Apr;23(2):e13560. doi: 10.1111/tid.13560. Epub 2021 Jan 16. PMID 33393172